CLINICAL TRIAL: NCT03855033
Title: Web-based High School Media Literacy for Healthy Relationships,
Brief Title: Feasibility Study of the Online High School Media Aware Program
Acronym: FS-OHSMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: iRT-Media Aware HS-Phase I
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Sexual Behavior
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Media Aware Sexual Health - High School (Experimental): Students received the web-based Media Aware Sexual Health - High School program.
  Interventions: Behavioral: Media Aware Sexual Health - High School
- Typical Health Education Programming (No Intervention): Students received their regular health education programming not related to sexual health education.

INTERVENTIONS:
Behavioral: Media Aware Sexual Health - High School — Media Aware Sexual Health is a web-based comprehensive sexual health education program for high school students that uses a media literacy approach.
  Other Names: Media Aware
  Arms: Media Aware Sexual Health - High School

SUMMARY:
This is a pretest-posttest feasibility study of Media Aware Sexual Health - High School, an interactive web-based comprehensive sexual health media literacy education program for high school students. The program is designed to develop students' critical thinking skills and promote sexual health. It is hypothesized that this program will enhance adolescents' media literacy skills, sexual health knowledge, cognitions (i.e., attitudes, self-efficacy, and norms), and behaviors regarding healthy sexual decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Students must be in grades 9 or 10 in participating classrooms at participating schools.
2. Students must be able to speak and read English because the study materials (e.g., questionnaires) and the program are in English.
3. Students must have appropriate permissions to receive sex education per school districts' policy (i.e., opt-in policy or opt-out policy).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 367 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Change in willingness to engage in unprotected sex | pretest and posttest (approximately one week after pretest)
  4-point Likert scale (strongly disagree; disagree; agree; strongly agree) assessing the degree to which one is willing to engage in unprotected sex (Suppose you were with a boyfriend/girlfriend. He/she wants to have sex, but neither of you have any form of protection. In this situation, how willing would you be to go ahead and hook-up anyway?).
Change in willingness to hook up against own wishes | pretest and posttest (approximately one week after pretest)
  4-point Likert scale (strongly disagree; disagree; agree; strongly agree) assessing the degree to which one is willing to hook up with someone even if they are not sure that they really want to. (Suppose you were with a boyfriend/girlfriend. He/she wants to hook-up, but you are not sure that you want to. In this situation, how willing would you be to go ahead and hook-up anyway?).
Change in intentions to use contraception/protection | pretest and posttest (approximately one week after pretest)
  4-point Likert scale (not at all likely; unlikely; likely; extremely likely) assessing intentions to use contraception (e.g., if you were to have vaginal or anal sex, how likely would you be to use a condom?).
Change in intentions to engage in sexual activity | pretest and posttest (approximately one week after pretest)
  4-point Likert scale (not at all likely; unlikely; likely; extremely likely) assessing participants intentions to engage in sex in the next year (How likely is that you will have any type of sexual contact with another person (oral sex, anal sex, vaginal sex, or genital-to-genital contact) in the next year?).

SECONDARY OUTCOMES:
Efficacy to refuse sexual activity | pretest and posttest (approximately one week after pretest)
  4-point Likert scale (strongly disagree; disagree; agree; strongly agree) assessing participants efficacy to refuse sex (e.g., I could say no to someone who is pressuring me to have sex).
Efficacy to communicate before sex | pretest and posttest (approximately one week after pretest)
  4-point Likert scale (strongly disagree; disagree; agree; strongly agree) assessing participants efficacy to communicate about sexual health (e.g., I could talk with a boy/girlfriend about using condoms for sexually transmitted infection protection).
Efficacy to use contraception/protection | pretest and posttest (approximately one week after pretest)
  4-point Likert scale (strongly disagree; disagree; agree; strongly agree) assessing participants efficacy to get and use contraception (e.g., If I wanted to, I could get condoms or another form of contraception).
Intentions to communicate before sex | pretest and posttest (approximately one week after pretest)
  4-point Likert scale (not at all likely; unlikely; likely; extremely likely) assessing intentions to communicate about sexual health before sex (e.g., Before deciding to have sex, how likely would you be to talk to a boy/girlfriend about HIV/AIDS or other sexually transmitted infections?).
Sexual health knowledge | pretest and posttest (approximately one week after pretest)
  Participants are asked several multiple choice and T/F questions about sexual health.
Norms - Frequency of teen risky sexual activity (%) | pretest and posttest (approximately one week after pretest)
  Participants are asked to indicate what percentage [0% = no teens; 100% = all teens] are engage in risky sexual activities (e.g., have sex with someone who is much older).
Norms - teen sexual activity (%) | pretest and posttest (approximately one week after pretest)
  Participants are asked to indicate what percentage [0% = no teens; 100% = all teens] are engage in sexual activity.
Perceived realism of media messages | pretest and posttest (approximately one week after pretest)
  Participants are asked on a 4-point Likert scale (strongly disagree; disagree; agree; strongly agree) the degree to which they agreed that teens on the media: 1) do things that average teens do; 2) act like average teens; 3) are as sexually experienced as average teens; 3) get pregnant as often as average teens; 4) get STIs as often as average teens.
Perceived similarity to media messages | pretest and posttest (approximately one week after pretest)
  Participants are asked on a 4-point Likert scale (strongly disagree; disagree; agree; strongly agree) the degree to which they agreed that: 1) The things I do in my life are similar to what I see teens do in the media; 2) I look like teens I see in the media; 3) I like the kinds of things that teens in the media like.
Cognitive elaboration of advertisement | pretest and posttest (approximately one week after pretest)
  Participants are shown an advertisement and responded on a 4-point Likert scale (not much at all; a little; a good amount; a lot) the extent to which they: 1) thought about the ad; 2) spent time thinking about the ad; and 3) paid attention to the ad.
Media Skepticism | pretest and posttest (approximately one week after pretest)
  Participants are asked on a 4-point Likert scale (strongly disagree; disagree; agree; strongly agree) the degree to which they agree with several statements about media (e.g., Media are dishonest about what happens when people drink alcohol).
Teen Sex Attitudes | pretest and posttest (approximately one week after pretest)
  Participants are asked on a 4-point Likert scale (strongly disagree; disagree; agree; strongly agree) the degree to which they agree with several statements about teen sex (e.g., it is ok for teens to be sexually active).
Risky Teen Sex Attitudes | pretest and posttest (approximately one week after pretest)
  Participants are asked on a 4-point Likert scale (strongly disagree; disagree; agree; strongly agree) the degree to which they agree with several statements about teens engaging in risky sexually behaviors (e.g., I believe it is ok for teens to do use alcohol or drugs before or during a sexual encounter.)
Teen Contraception Use Attitudes | pretest and posttest (approximately one week after pretest)
  Participants are asked on a 4-point Likert scale (strongly disagree; disagree; agree; strongly agree) the degree to which they agree with several statements about teen contraception use (e.g., I believe if a teen is going to have sex, they should always use a condom.)
Teen Sexual Communication Attitudes | pretest and posttest (approximately one week after pretest)
  Participants are asked on a 4-point Likert scale (strongly disagree; disagree; agree; strongly agree) the degree to which they agree with several statements about teen sexual communication (e.g., Before deciding to have sex, I believe teens should talk with their parents or another trusted adult).

OTHER OUTCOMES:
Intent to intervene as bystander | pretest and posttest (approximately one week after pretest)
  Participants are asked on a 4-point Likert scale (not likely at all; Unlikely; Likely; Extremely likely) how likely they would be to intervene as a bystander (e.g., Approach a friend if I thought they were in an abusive relationship and let them know that I am here to help)
Efficacy to intervene as bystander | pretest and posttest (approximately one week after pretest)
  Participants are asked to indicate on a scale on 0 (Can't do) to 100 (Very Certain) their degree of confidence in several behaviors (e.g., I could talk to a friend who I suspected is in an abusive relationship.)
Belief in rape myths | pretest and posttest (approximately one week after pretest)
  Participants are asked on a 4-point Likert scale (strongly disagree; disagree; agree; strongly agree) their level of agreement on several items pertaining to myths about rape (e.g., It shouldn't be considered rape if a guy is drunk and didn't realize what he was doing.)
Acceptance of strict gender role stereotypes | pretest and posttest (approximately one week after pretest)
  Participants are asked on a 4-point Likert scale (strongly disagree; disagree; agree; strongly agree) their level of agreement on several items pertaining to strict gender role stereotypes (e.g., Raising children is primarily a woman's responsibility).
Acceptance of dating violence | pretest and posttest (approximately one week after pretest)
  Participants are asked on a 4-point Likert scale (strongly disagree; disagree; agree; strongly agree) their level of agreement on several items pertaining to dating violence (e.g., It is okay for people to hit their girlfriends/boyfriends if they did something to make them mad).

CONTACTS AND LOCATIONS:
Locations (1):
- innovation Research & Training, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No